CLINICAL TRIAL: NCT00377169
Title: Genomics: A Substudy of a Large, Simple Trial Comparing Two Strategies for Management of Anti-Retroviral Therapy (The SMART Study)
Brief Title: Collection of Blood Samples From SMART Study Participants for Future Genetic Studies
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Community Programs for Clinical Research on AIDS (Network)
Other Study IDs: CPCRA 065H; SMART
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2006-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to collect blood samples from SMART study participants to use in future genetic studies.

DETAILED DESCRIPTION:
Despite progress in the treatment of HIV and a greater understanding of the pathophysiology of HIV infection, there are still unexplained differences in both the progression of untreated HIV infection and response to antiretroviral therapy. These differences are likely related to the unique genetic makeup of individuals with HIV infection. Particular genes may offer protection against HIV infection, while other genes may make disease progression more likely. Knowing more about the genetic makeup of HIV infected individuals may lead to the development of a targeted treatment strategy based on an individual's specific risk of disease progression and sensitivity to medication toxicity. The purpose of this substudy is to collect blood samples from SMART study participants. The samples will be used in future Community Programs for Clinical Research on AIDS (CPCRA) studies investigating the link between human genetic factors and clinical outcome data.

This study will enroll individuals currently participating in the SMART study. Participants will provide one blood sample. Individual test results from future blood analyses will not be provided to a patient unless they may have profound health implications for that patient.

ELIGIBILITY:
Inclusion Criteria:

* Coenrollment in the SMART study
* Parent or guardian willing to provide informed consent, if applicable

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3261 (Estimated)
Dates: Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Uy, MD, Study Chair — AIDS Research Alliance Chicago (ARAC), University of Illinois at Chicago; Roberto Arduino, MD, Study Chair — The University of Texas Health Science Center, Houston; Fraser Drummond, MBChB, MRCA, DA (UK), Study Chair — National Centre in HIV Epidemiology and Clinical Research, University of New South Wales; Daniela Gey, MD, Study Chair — Copenhagen HIV Programme, Hvidovre University Hospital; Adrian Palfreeman, MD, Study Chair — Peterborough and Stamford Hospitals NHS Foundation Trust
Locations (42):
- United States (17):
  - AltaMed Health Services Corporation, Los Angeles, California
  - Los Angeles Gay & Lesbian Community Service Center, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - VA Greater Loss Angeles Healthcare System, Los Angeles, California
  - Comprehensive Care Center/North Broward Hospital, Fort Lauderdale, Florida
  - Hillsborough County Health Department, Tampa, Florida
  - Absolute Care Clinic, Atlanta, Georgia
  - AID Atlanta/Morehouse Medical School Ryan White Cl, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta (ARCA) Central, Atlanta, Georgia
  - Dr. Dennis Melton (private practice), Atlanta, Georgia
  - Dr. Melanie Thompson and Dr. Annette Bernard (private practice), Atlanta, Georgia
  - Dr. Richard Hudson (private practice), Atlanta, Georgia
  - Mayo Clinic/CORNET, Rochester, Minnesota
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Westchester Medical Center/New York Medical College, Valhalla, New York
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Froedtert and Medical College I.D. Clinic, Milwaukee, Wisconsin
- Gladstone Road Medical Centre, Highgate Hill, American Samoa
- Australia (3):
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth
  - Westmead Hospital, Westmead
- C.H.U. St. Pierre Center Hospitalier Universitaire, Brussels, Belgium
- Clinique Medicale L'actuel, Montreal, Quebec, Canada
- Fundacion Arriaran Santa Elvira, Santiago, Chile
- Arbus Universitetshospital, Skejby Department of Infectious Diseases, Brendstrupgaardvej Aarhus, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- Germany (4):
  - University Hospital Koln (Cologne), Cologne
  - J.W. Goethe University Hospital, Frankfurt
  - ifi Institut, Hamburg
  - Infektionsambulanz und Tagesklinik Poliklinik Innenstadt der, Munich
- AIDS Medical Center, International Medical Center, Tokyo, Japan
- University Hospital Center Ibn Rochd, Casablanca, Morocco
- New Zealand (3):
  - Wellington Hospital, Newtown, Wellington Region
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Wroclaw University School of Medicine, Koszarawa, Poland
- Portugal (3):
  - Centro Hospital de Cascais, Cascais
  - Hospital de Santa Maria, Lisbon
  - Hospital Joaquim Urbano, Porto
- The Gambia (2):
  - Medizinische Universitatsklinik, Bonn
  - Klinikum der Ruprecht-Karis-Universitat (U. Hospit), Heidelberg
- Catedra de Enfermedades Infecciosas, Montevideo, Uruguay

REFERENCES:
- See also: Click here for more information on CPCRA 065 — http://clinicaltrials.gov/show/NCT00027352